CLINICAL TRIAL: NCT02184351
Title: A Prospective Randomized, Blinded Parallel Group Study of Clotrimazole Troches vs. Mycelex® Troches (10 mg Troche Five Times a Day for 14 Days) in Patients With Human Insufficiency Virus (HIV) Infection for the Treatment of Oropharyngeal Candidiasis
Brief Title: Clotrimazole vs. Mycelex® in Patients With Human Insufficiency Virus (HIV) Infection for the Treatment of Oropharyngeal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1190.1
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral

ARMS (2):
- Roxanes's clotrimazole troches (Experimental)
  Interventions: Drug: Roxanes's clotrimazole troches
- Mycelex® troches (Active Comparator)
  Interventions: Drug: Mycelex® troches

INTERVENTIONS:
Drug: Roxanes's clotrimazole troches
  Arms: Roxanes's clotrimazole troches
Drug: Mycelex® troches
  Arms: Mycelex® troches

SUMMARY:
The objectives of this study are to compare the efficacy and safety of Roxane's clotrimazole troches vs. Mycelex troches in HIV positive patients with oropharyngeal candidiasis, where this condition has been diagnosed by clinical examination and confirmed by fungal culture.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV positive status
* Clinical examination of oropharynx is consistent with diagnosis of oral Candidiasis (such as creamy, white, curdlike patches or erythematous lesions on mucosal surfaces)
* Findings on direct microscopic examination (Gram Stain or potassium hydroxide smear) consistent with Candida species or positive fungal culture for Candida species, with culture obtained in the 2 days preceding initiation of therapy with the study drug
* Male or female patients ≥ 18 years
* For women of childbearing potential: negative blood or urine pregnancy test and agreement to use adequate contraception (investigator's discretion) while on study drug
* Mental status allows comprehension of instructions for troche administration
* Written informed consent

Exclusion Criteria:

* Sings of symptoms suggestive of esophageal Candidiasis (such as dysphagia or odynophagia) unless the results of an endoscopic evaluation of the esophagus are negative
* Presence of perioral lesions only
* Use of other antifungal agents within 5 days of enrollment to the study
* Pregnant or lactating women
* History of hypersensitivity to imidazole or azole compounds
* Patient unwilling or unable to be followed at the study center for the duration of the study (3 weeks)
* Patients has received an investigational drug in the last 30 days
* Treatment with another investigational drug is planned within the next 3 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2001-05; Primary Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Percent of patients that have a clinical response assessed by symptoms and physical examination | Day 21

SECONDARY OUTCOMES:
Incidence of negative fungal cultures of the oropharynx for Candida species | 7 days after end of treatment
Incidence of negative fungal cultures of the oropharynx for Candida species | after 14 days of treatment
Clinical response by symptom assessment and physical examination | after 7 and 14 days of treatment
Assessment of compliance with Treatment by troche Count and Patient interview | after 7 and 14 days of treatment